CLINICAL TRIAL: NCT02207608
Title: Pilot Study of Influence of Hyaluronic Acid (HA) on Bacillus Calmette-Guérin (BCG) Local Side Effects
Brief Title: Influence of Hyaluronic Acid on Bacillus Calmette-Guérin Local Side Effects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Enrico Finazzi Agro, Associate Professor, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA-1
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Results first posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Poisoning by BCG Vaccine
Keywords: BCG; hyaluronic acid; non-muscle invasive bladder cancer; non bacterial cystitis
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BCG alone (Immucist®) (Active Comparator): Group A receive BCG (Immucist® 81 mg, Sanofi-Aventis Group) alone
  Interventions: Drug: BCG (Immucist®)
- Hyaluronic acid (Experimental): Group B receive BCG and HA 40 mg (Cystistat, Mylan, Pittsburgh, PA, U.S.A.).
  Interventions: Drug: Hyaluronic Acid; Drug: BCG (Immucist®)

INTERVENTIONS:
Drug: Hyaluronic Acid — Add hyaluronic acid to BCG Treatment
  Other Names: Cystistat (Mylan, Pittsburgh, PA, U.S.A.)
  Arms: Hyaluronic acid
Drug: BCG (Immucist®) — Usual BCG treatment
  Other Names: BCG

SUMMARY:
The purpose of this study is to evaluate a possible role of intravesical Hyaluronic Acid in reducing local toxicity of Bacillus Calmette Guerin (BCG) used to treat bladder urothelial cell carcinoma.

DETAILED DESCRIPTION:
Bacillus Calmette-Guérin (BCG) is considered the most effective treatment to increase disease-free interval and reduce progression of non-muscle invasive bladder cancer (NMIBC) [1]. Although considered safe, BCG can produce both local and systemic side effects leading to treatment discontinuation or interruption. The most common local side-effects of BCG intravesical instillations include cystitis, characterized by irritative voiding symptoms and hematuria, which occur in approximately 75% of all patients. More rarely, serious local adverse events as a result of BCG infection, such as symptomatic granulomatous prostatitis and epididymo-orchitis, might occur and require permanent discontinuation of BCG treatment. Systemic side-effects include flu-like symptoms, such as general malaise and fever, occuring in approximately 40% of patients. A high persistent fever might be related to BCG infection or sepsis. Local and systemic side-effects might lead to discontinue intravesical BCG treatment in approximately 20% of patients [2]. Up to 54% of the patients undergoing intravesical therapy with chemotherapeutic agents to treat superficial bladder tumours can be affected by nonbacterial cystitis [3].

Several solutions have been proposed to reduce the occurrence of side effects from BCG with the aim to limit BCG discontinuation and the concomitant discomfort during endovesical treatment. Some Authors have proposed to avoid BCG administration in case of TUR within previous 2 weeks, traumatic catheterization, macroscopic hematuria, urethral stenosis, active tuberculosis, prior Bacillus Calmette-Guérin sepsis, immuno-suppression or urinary tract infection [4]. Other procedures include the prophylactic administration of isoniazid [5] or ofloxacin [6,7] or usually involve BCG dose reductions [8]. In common practice antimicrobials, anticholinergics, anaesthetics and analgesics are often used to relieve patients' symptoms.

Glycosaminoglycan (GAG) substitution therapy is an emerging treatment of Bladder Pain Syndrome/Interstitial Cystitis (BPS/IC) and response rates between 30% and 80% have been described with intravesical administration of various GAGs (hyaluronic acid, pentosan polysulfate, heparin, chondroitin sulfate, and dimethyl sulfoxide) [9,10]. Few papers report the results of GAG substitution therapy in the treatment of radiation and chemical cystitis [9,10]. To our knowledge, to date, only two papers have described GAG use in the treatment of BCG local side effects; this papers show very good results, with significant reduction of lower urinary tract symptoms after intravesical administration of HA [11,12].

Aim of the present randomized pilot study was to evaluate if the sequential administration of HA and BCG could be safe in prevention of early recurrence and progression of bladder tumor, and safe in reduction of local side-effects in patients with high risk NMIBC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven non-muscle invasive bladder cancer;
* Indication to intravesical instillation of BCG according to EAU guidelines;
* Age > 18 years;
* Willingness, to participate to the study;
* Written informed consent.

Exclusion Criteria:

* Previous or ongoing BCG or different intravesical instillations;
* Urinary tract infections (UTI) or other known pathologies of the lower urinary tract;
* Indication for a radical cystectomy;
* Severe systemic disorders, including neurological pathologies, kidney, liver or heart failure;
* Contraindications to BCG use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

REFERENCES:
- [Derived] Topazio L, Miano R, Maurelli V, Gaziev G, Gacci M, Iacovelli V, Finazzi-Agro E. Could hyaluronic acid (HA) reduce Bacillus Calmette-Guerin (BCG) local side effects? Results of a pilot study. BMC Urol. 2014 Aug 13;14:64. doi: 10.1186/1471-2490-14-64. PMID 25123116

RESULTS

PARTICIPANT FLOW:
Groups:
- BCG Alone (Immucist®): Group A receive BCG (Immucist® 81 mg, Sanofi-Aventis Group) alone
  BCG (Immucist®)
- Hyaluronic Acid: Group B receive BCG and HA 40 mg (Cystistat, Mylan, Pittsburgh, PA, U.S.A.).
  Hyaluronic Acid
  BCG (Immucist®)
Period: Overall Study
Arm/Group | BCG Alone (Immucist®) | Hyaluronic Acid
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BCG Alone (Immucist®) | Hyaluronic Acid | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Mean (Full Range); unit: years] | 66 [60 to 81] | 68 [54 to 75] | 67 [54 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 11 | 11 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 15 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale for Pain
Description: 1 to 10 scale (1 minimum pain perceivable; 10 unbearable pain, as perceived by the patient)
Time Frame: Before and after six weeks of treatment (end of induction course)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BCG Alone (Immucist®) | Hyaluronic Acid
Number analyzed (Participants) | 14 | 15
units on a scale
  Data Before treatment | 4.5 (2) | 4.9 (1.8)
  Data after treatment | 5.8 (1) | 4.2 (1.6)

ADVERSE EVENTS:
Arm/Group | BCG Alone (Immucist®) | Hyaluronic Acid
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCG Alone (Immucist®) (N=15) | Hyaluronic Acid (N=15)
Urgency (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No